## Medication Dispensing System to Support Medication Adherence for Individuals Living at Home with Chronic Conditions: A Randomized Controlled Trial

NCT04339296

Ethics ID: PRO 00087782

November 10, 2019

Descriptive and inferential statistics was used to compare baseline characteristics and adherence among the intervention and control groups. For the baseline, investigators compared the characteristic between the intervention and control group. A Chi-square test of independence was used for categorical variables such as gender, ethnicity, and medication management method. An independent sample t-test was performed for continuous variables such as age, number of chronic conditions, number of medications and medication adherence. Pairwise comparison was completed for self-reported health status, medication management and adherence scores at baseline (pretest) and six month (posttest). Intention-to-treat (ITT) analysis was utilized to keep all of participant's data in the group they were originally assigned by the randomization process. Statistical tests for inferential statistics was set at 95% confidence level. All the data was entered and analyzed using SPSS Statistics version 25.

<sup>1</sup> McCoy CE. Understanding the intention-to-treat principle in randomized controlled trials. Western Journal of Emergency Medicine. 2017 Oct;18(6):1075-1078.